CLINICAL TRIAL: NCT02737267
Title: Development of a Nutrigenetic Test for Personalized Prescription of Body Weight Loss Diets (Obekit)
Acronym: Obekit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 132/2015
Record Dates: First submitted 2016-03-10; First posted 2016-04-13 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2015-11

CONDITIONS: Body Weight Changes
Keywords: Genetics; Polymorphism; Epigenetics; Metagenomics; Metabolomics; Metabolic syndrome conditions; Precision nutrition
MeSH Terms: conditions — Body Weight Changes | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderately high protein diet (Experimental): Caloric restriction (-30% total energy intake) Macronutrient distribution: 40% of the energy derived from carbohydrates, 30% of the energy derived from protein and 30% of the energy derived from fat
  Interventions: Behavioral: Moderately high protein diet
- Low fat diet (Placebo Comparator): Caloric restriction (-30% total energy intake) Macronutrient distribution: 60% of the energy derived from carbohydrates, 18% of the energy derived from protein and 22% of the energy derived from fat
  Interventions: Behavioral: Low fat diet

INTERVENTIONS:
Behavioral: Moderately high protein diet — After the recruitment randomization of the study participants, the study will consists of a 4-month nutritional intervention ("body weight loss period") followed by a second 6-month period ("body weight maintenance period") in which the subjects of the study will continue with the assigned diet, but without any energy restriction.
  Arms: Moderately high protein diet
Behavioral: Low fat diet — After the recruitment randomization of the study participants, the study will consists of a 4-month nutritional intervention ("body weight loss period") followed by a second 6-month period ("body weight maintenance period") in which the subjects of the study will continue with the assigned diet, but without any energy restriction.the energy derived from fat
  Arms: Low fat diet

SUMMARY:
This study evaluates the relationship between several genetic variants and the response to a hypocaloric diet, in order to design a genetic test which permits prescribe the more personalized diet for each individual according to her genotype. Half of the participants will assigned to a moderate high protein diet, while the other half will assigned to a high carbohydrate diet.

DETAILED DESCRIPTION:
Obesity has reached epidemic proportions becoming a major global public health challenge since it is associated with an increased risk of type 2 diabetes, cardiovascular disease, stroke, arthritis and some forms of cancer. Therefore, a large number of strategies have been investigated in order to induce a negative energy balance and consequently body weight loss mainly inducing a low calorie diet and sometimes accompanied by an increase in physical activity. However, individual responses to body weight loss interventions vary widely and several studies have aimed to identify psychological, behavioral and personal predictors of this variability.

In this context, the hypothesis of the present study is that part of the interindividual variability in relation to the success of certain weight loss treatments is based on gene-diet interactions. Depending on the composition of the diet and the genotype of each individual, it is more or less easy to reduce and maintenance body weight.

After the recruitment and selection of the study participants, the study will consists of a 4-month hypocaloric diet ("body weight loss period") followed by a second 6-month period ("body weight maintenance period") in which the subjects of the study will continue with the diet, but without any energy restriction. The participants will assigned to one of the two hypocaloric diets (-30% of the studied requirements for each individual) with different macronutrient composition:

* Moderately high protein diet: 40% of the energy derived from carbohydrates, 30% of the energy derived from protein and 30% of the energy derived from fat.
* Low fat diet: 60% of the energy derived from carbohydrates, 30% of the energy derived from protein and 30% of the energy derived from fat.

A group of normal weight individuals (n 12) will be recruited in order to compare the different parameters obtained in the obese subjects with those of normal population. They will be not subjected to any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 25 and 40 kg/m2
* Physical examination and vital signs normal, or is considered abnormal, but clinically insignificant by researcher.
* In the case of individuals with chronic stable dose drug treatment and during the last 3 previous months at baseline, the investigator will assess their possible inclusion.

Exclusion Criteria:

* BMI less than 25 or higher than 40 kg/m2
* Pregnant women
* Breastfeeding period. If artificial feeding until 6 months after birth.
* Type 1 diabetes
* Severe kidney diseases
* Severe digestive system diseases
* Electrolyte disorders (disorders of sodium, potassium, calcium, chlorine, phosphorus, magnesium)
* Acute cardiovascular diseases
* Cancer
* Anemia
* Eating disorders
* Recent prescription drug treatment (without stable doses scheduled)
* Drug therapy that can influence weight loss as corticosteroids.
* Some type of cognitive impairment and / psychic
* Subjects in which poor collaboration or, in the investigator's opinion, have difficulty following the procedures of the study is foreseen
* Lack of commitment (at the discretion of the investigator) with the intervention, suspected non-compliance, or real difficulties to follow the development of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in body weight at Week 16 | Baseline and 16 Weeks
Change in body weight at Week 40 | 16 Weeks and 40 Weeks

SECONDARY OUTCOMES:
Height | Baseline
Change in waist and hip circumferences at 16 Weeks | Baseline and 16 Weeks
  Waist and hip circumferences will be measured with a tape measure at baseline and at the end of the body weight loss period (16 weeks)
Change in waist and hip circumferences at 40 Weeks | 16 Weeks and 40 Weeks
  Waist and hip circumferences will be measured with a tape measure at the end of the body weight loss period (16 weeks) and at the end of the body weight maintenance period (40 Weeks)
Change in body fat mass at 16 Weeks | Baseline and 16 Weeks
  Fat mass will be measured by bioelectric bioimpedance and Dual X-ray absorptiometry at baseline and at the end of the body weight loss period (16 Weeks)
Change in body fat mass at 40 Weeks | 16 Weeks and 40 Weeks
  Fat mass will be measured by bioelectric bioimpedance and Dual X-ray absorptiometry at the end of the body weight loss period (16 weeks) and at the end of the body weight maintenance period (40 Weeks)
Single nucleotide polymorphisms (SNPs) | Baseline
  Single nucleotide polymorphisms will be measured from Genomic DNA from oral epithelial cells (collected in ORAcollect DNA, DNAGenotek) and from peripheral blood mononuclear cells (PBMC) by using massive sequencing in a Ion Torrent sequencer
Changes in DNA methylation levels at 16 Weeks | Baseline and 16 Weeks
  DNA methylation levels will be measured in PBMC by Microarray (Illumina. 450k methylation array) and validation specific sites by Sequenom (MassArray) and Methylationsensitive High-Resolution Melting (MS-HRM) (Real Time PCR) at baseline and at the end of the body weight loss period (16 Weeks)
Changes in DNA methylation levels at 40 Weeks | 16 Weeks and 40 Weeks
  DNA methylation levels will be measured in PBMC by Microarray (Illumina 450k methylation array) and validation specific sites by Sequenom (MassArray) and MS-HRM (Real Time PCR) at the end of the body weight loss period (16 weeks) and at the end of the maintenance body weight period (40 Weeks)
Changes in metabolic profiling at 16 Weeks | Baseline and 16 Weeks
  Metabolic profiling will be measured in urine by High Performance Liquid Chromatography-Mass Spectrometry (HPLC-MS) at baseline and at the end of the body weight loss period (16 Weeks)
Changes in metabolomic profile at 40 Weeks | 16 Weeks and 40 Weeks
  Metabolomic profile will be measured in urine by HPLC-MS at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in lipidomic profile at 16 Weeks | Baseline and 16 Weeks
  Lipidomic profile will be measured in plasma by HPLC-MS at baseline and at the end of the body weight loss period (16 Weeks)
Changes in lipidomic profile at 40 Weeks | 16 Weeks and 40 Weeks
  Lipidomic profile will be measured in plasma by HPLC-MS at the end of the body weight loss period (16 weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in proteomic profile at 16 Weeks | Baseline and 16 Weeks
  Proteomic profile will be measured in plasma by Two-Dimensional Fluorescence Difference Gel Electrophoresis (2D-DIGE) and Liquid Chromatography Electrospray Ionization with Tandem Mass Spectrometry (LC-ESI-MS/MS) at baseline and at the end of the body weight loss period (16 Weeks)
Changes in proteomic profile at 40 Weeks | 16 Weeks and 40 Weeks
  Proteomic profile will be measured in plasma by 2D-DIGE and LC-ESI-MS/MS at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in gut microbiota composition at 16 Weeks | Baseline and 16 Weeks
  Gut microbiota composition will be measured by Pyrosequencing 16SR RNA at baseline and at the end of the body weight loss period (16 Weeks)
Changes in gut microbiota composition at 40 Weeks | 16 Weeks and 40 Weeks
  Gut microbiota composition will be measured by Pyrosequencing 16SR RNA at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in messenger ribonucleic acid (mRNA) expression at 16 Weeks | Baseline and 16 Weeks
  mRNA expression will be measured by GeneChip Human Transcriptome Array 2.0 (Affimetrix) at baseline and at the end of the body weight loss period (16 Weeks)
Changes in mRNA expression at 40 Weeks | 16 Weeks and 40 Weeks
  mRNA expression will be measured by GeneChip Human Transcriptome Array 2.0 (Affimetrix) at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in microARNs in exosomes at 16 weeks | Baseline and 16 Weeks
  microARNs levels in exosomes will be measured by NGS Illumina Myseq at baseline and at the end of the body weight loss period (16 Weeks)
Changes in microARNs in exosomes at 40 weeks | 16 Weeks and 40 Weeks
  microARNs levels in exosomes will be measured by next-generation sequencing (NGS) Illumina Myseq at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in DNA oxidation at 16 weeks | Baseline and 16 Weeks
  DNA oxidation will be measured by 8-hydroxy-deoxyguanosine at baseline and at the end of the body weight loss period (16 Weeks)
Changes in DNA oxidation at 40 weeks | 16 Weeks and 40 Weeks
  DNA oxidation will be measured by 8-hydroxy-deoxyguanosine at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in serum glucose levels at 16 Weeks | Baseline and 16 weeks
  Serum glucose levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in serum glucose levels at 40 Weeks | 16 Weeks and 40 Weeks
  Serum glucose levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in serum insulin concentration at 16 Weeks | Baseline and 16 Weeks
  Serum insulin concentration will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in serum insulin concentration at 40 Weeks | 16 Weeks and 40 Weeks
  Serum insulin concentration will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in serum lipid metabolism markers at 16 Weeks | Baseline and 16 Weeks
  Serum free fatty acids, triglycerides, total cholesterol, LDL cholesterol and HDL cholesterol concentrations will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in serum lipid metabolism markers at 40 Weeks | 16 Weeks and 40 Weeks
  Serum free fatty acids, triglycerides, total cholesterol, LDL cholesterol and HDL cholesterol concentrations will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in serum total protein concentration at 16 Weeks | Baseline and 16 Weeks
  Serum total protein concentration will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in serum total protein concentration at 40 Weeks | 16 Weeks and 40 Weeks
  Serum total protein concentration will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in serum uric acid levels at 16 Weeks | Baseline and 16 Weeks
  Serum uric acid levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in serum uric acid levels at 40 Weeks | 16 Weeks and 40 Weeks
  Serum uric acid levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in serum transaminases concentrations at 16 Weeks | Baseline and 16 Weeks
  Serum transaminases (AST & ALT) concentrations will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in serum transaminases concentrations at 40 Weeks | 16 Weeks and 40 Weeks
  Serum transaminases (AST & ALT) concentrations will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in serum homocystein concentration at 16 Weeks | Baseline and 16 Weeks
  Serum homocystein concentration will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in serum homocystein concentration at 40 Weeks | 16 Weeks and 40 Weeks
  Serum homocystein concentration will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in vascular endothelial growth factor (VEGF) at 16 Weeks | Baseline and 16 Weeks
  VEGF levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in vascular endothelial growth factor (VEGF) at 40 Weeks | 16 Weeks and 40 Weeks
  VEGF levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in asymmetric dimethylarginine (ADMA) at 16 Weeks | Baseline and 16 Weeks
  ADMA levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in asymmetric dimethylarginine (ADMA) at 40 Weeks | 16 Weeks and 40 Weeks
  ADMA levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in PAI-1 concentration at 16 Weeks | Baseline and 16 Weeks
  PAI-1 concentration will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in plasminogen activator inhibitor-1 (PAI-1) concentration at 40 Weeks | 16 Weeks and 40 Weeks
  PAI-1 concentration will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in nitric oxide levels at 16 Weeks | Baseline and 16 Weeks
  Nitric oxide levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in nitric oxide levels at 40 Weeks | 16 Weeks and 40 Weeks
  Nitric oxide levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in blood pressure at 16 Weeks | Baseline and 16 Weeks
  Changes in diastolic and systolic blood pressure will be measured at baseline and at the end of the body weight loss period (16 Weeks)
Changes in blood pressure at 40 Weeks | 16 Weeks and 40 Weeks
  Changes in diastolic and systolic blood pressure will be measured at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in plasma C-Reactive Protein levels at 16 Weeks | Baseline and 16 Weeks
  C-Reactive Protein levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in plasma C-Reactive Protein levels at 40 Weeks | 16 Weeks and 40 Weeks
  C-Reactive Protein levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in plasma interleukin-6 (IL-6) and interleukin-10 (IL-10) levels at 16 Weeks | Baseline and 16 Weeks
  IL-6 and IL-10 levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in plasma IL-6 and IL-10 levels at 40 Weeks | 16 Weeks and 40 Weeks
  IL-6 and IL-10 levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in plasma tumor necrosis factor-alpha (TNF-alpha) levels at 16 Weeks | Baseline and 16 Weeks
  TNF-alpha levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in plasma TNF-alpha levels at 40 Weeks | 16 Weeks and 40 Weeks
  TNF-alpha levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in adiponectin levels at 16 Weeks | Baseline and 16 Weeks
  Adiponectin levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in adiponectin levels at 40 Weeks | 16 Weeks and 40 Weeks
  Adiponectin levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in chemerin levels at 16 Weeks | Baseline and 16 Weeks
  Chemerin levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in chemerin levels at 40 Weeks | 16 Weeks and 40 Weeks
  Chemerin levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in leptin levels at 16 Weeks | Baseline and 16 Weeks
  Leptin levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in leptin levels at 40 Weeks | 16 Weeks and 40 Weeks
  Leptin levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in apelin levels at 16 Weeks | Baseline and 16 Weeks
  Apelin levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in apelin levels at 40 Weeks | 16 Weeks and 40 Weeks
  Apelin levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in haptoglobin levels at 16 Weeks | Baseline and 16 Weeks
  Haptoglobin levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in haptoglobin levels at 40 Weeks | 16 Weeks and 40 Weeks
  Haptoglobin levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in amyloid A levels at 16 Weeks | Baseline and 16 Weeks
  Amyloid A levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in amyloid A levels at 40 Weeks | 16 Weeks and 40 Weeks
  Amyloid A levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in leukocytes levels at 16 Weeks | Baseline and 16 Weeks
  Leukocytes levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in leukocytes levels at 40 Weeks | 16 Weeks and 40 Weeks
  Leukocytes levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in plasma LDL-ox levels at 16 Weeks | Baseline and 16 Weeks
  Levels of LDL-ox in plasma will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in plasma LDL-ox levels at 40 Weeks | 16 Weeks and 40 Weeks
  Levels of LDL-ox in plasma will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in glutathione peroxidase activity at 16 Weeks | Baseline and 16 Weeks
  Glutathione peroxidase activity will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in glutathione peroxidase activity at 40 Weeks | 16 Weeks and 40 Weeks
  Glutathione peroxidase activity will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in reduced and oxidized glutathione levels at 16 Weeks | Baseline and 16 Weeks
  Reduced and oxidized glutathione levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in reduced and oxidized glutathione levels at 40 Weeks | 16 Weeks and 40 Weeks
  Reduced and oxidized glutathione levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in superoxide dismutase levels at 16 Weeks | Baseline ant 16 Weeks
  Superoxide dismutase levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in superoxide dismutase levels at 40 Weeks | 16 Weeks and 40 Weeks
  Superoxide dismutase levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in serum isoprostanes levels at 16 Weeks | Baseline and 16 Weeks
  Serum isoprostanes levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in serum isoprostanes levels at 40 Weeks | 16 Weeks and 40 Weeks
  Serum isoprostanes levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in plasma malonyldialdehyde (MDA) concentration at 16 Weeks | Baseline and 16 Weeks
  MDA concentration will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in plasma malonyldialdehyde (MDA) concentration at 40 Weeks | 16 Weeks and 40 Weeks
  MDA concentration will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in monoamines levels at 16 Weeks | Baseline and 16 Weeks
  Plasma monoamines (dopamine, dopac, homovalic acid, serotonin, noradrenalin) levels will be measured in a fasting state at baseline and at the end of the body weight loss period (16 Weeks)
Changes in monoamines levels at 40 Weeks | 16 Weeks and 40 Weeks
  Plasma monoamines (dopamine, dopac, homovalic acid, serotonin, noradrenalin) levels will be measured in a fasting state at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in physical activity at 16 Weeks | Baseline and 16 Weeks
  Physical activity level will be measured by a validated physical activity questionnaire and by a pedometer at baseline and at the end of the body weight loss period (16 Weeks)
Changes in physical activity at 40 Weeks | 16 Weeks and 40 Weeks
  Physical activity level will be measured by a validated physical activity questionnaire and by a pedometer at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in depression degree at 16 Weeks | Baseline and 16 Weeks
  Depression degree will be measured by the Beck Depression Inventory at baseline and at the end of the body weight loss period (16 Weeks)
Changes in depression degree at 40 Weeks | 16 Weeks and 40 Weeks
  Depression degree will be measured by the Beck Depression Inventory at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in anxiety degree at 16 Weeks | Baseline and 16 Weeks
  Anxiety degree will be measured by the State-Trait Anxiety Inventory (STAI) at baseline and at the end of the body weight loss period (16 Weeks)
Changes in anxiety degree at 40 Weeks | 16 Weeks and 40 Weeks
  Anxiety degree will be measured by the State-Trait Anxiety Inventory (STAI) at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in the chronotype at 16 Weeks | Baseline and 16 Weeks
  Chronotype will be defined by two questionnaires at baseline and at the end of the intervention period (16 Weeks)
Changes in the chronotype at 40 Weeks | 16 Weeks and 40 Weeks
  Chronotype will be defined by two questionnaires at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)
Changes in food intake at 16 Weeks | Baseline and 16 weeks
  Food intake will be evaluated by a 72 hours dietary record at baseline and at the end of the body weight loss period (16 Weeks)
Changes in food intake at 40 Weeks | Baseline and 40 weeks
  Food intake will be evaluated by a 72 hours dietary record and by a validated Food Frequency Questionnaire at baseline and at the end of the body weight maintenance period (40 Weeks)
Changes in satiety at 16 Weeks | Baseline and 16 Weeks
  Satiety will be evaluated by the Visual Analogue Scale (VAS) at baseline and at the end of the body weight loss period (16 Weeks)
Changes in satiety at 40 Weeks | 16 Weeks and 40 Weeks
  Satiety will be evaluated by the Visual Analogue Scale (VAS) at the end of the body weight loss period (16 Weeks) and at the end of the body weight maintenance period (40 Weeks)

CONTACTS AND LOCATIONS:
Overall Officials: J. Alfredo Martínez, MD, PhD, Principal Investigator — Centre for Nutrition Research, University of Navarra. CIBER Obesity and Physiopathology of Nutrition (CIBERobn), Institute of Health Carlos III Madrid Spain; Fernando J. Corrales, PhD, Principal Investigator — CIMA, University of Navarra; Femín I Milagro, PhD, Study Chair — Centre for Nutrition Research, University of Navarra. CIBER Obesity and Physiopathology of Nutrition (CIBERobn), Institute of Health Carlos III Madrid Spain; Jose Ignacio Riezu, PhD, Study Chair — Centre for Nutrition Research, University of Navarra; Carlos González-Navarro, PhD, Study Chair — Centre for Nutrition Research, University of Navarra; Marta Cuervo, PhD, Study Chair — Centre for Nutrition Research, University of Navarra; Iosune Zubieta, Study Chair — Centre for Nutrition Research, University of Navarra; Blanca Esther Martínez de Morentin, MD, Study Chair — Centre for Nutrition Research, University of Navarra; Leticia Goñi, Study Chair — Centre for Nutrition Research, University of Navarra; Santiago Navas, PhD, Study Chair — Centre for Nutrition Research, University of Navarra. CIBER Obesity and Physiopathology of Nutrition (CIBERobn), Institute of Health Carlos III Madrid Spain
Locations (1):
- Centre for Nutrition Research, University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Alvarez NC, Riezu-Boj JI, Martinez JA, Garcia-Calzon S, Milagro FI. A Predictive Tool Based on DNA Methylation Data for Personalized Weight Loss through Different Dietary Strategies: A Pilot Study. Nutrients. 2023 Dec 6;15(24):5023. doi: 10.3390/nu15245023. PMID 38140282
- [Derived] Cuevas-Sierra A, Milagro FI, Guruceaga E, Cuervo M, Goni L, Garcia-Granero M, Martinez JA, Riezu-Boj JI. A weight-loss model based on baseline microbiota and genetic scores for selection of dietary treatments in overweight and obese population. Clin Nutr. 2022 Aug;41(8):1712-1723. doi: 10.1016/j.clnu.2022.06.008. Epub 2022 Jun 16. PMID 35777110
- [Derived] Cuevas-Sierra A, Romo-Hualde A, Aranaz P, Goni L, Cuervo M, Martinez JA, Milagro FI, Riezu-Boj JI. Diet- and sex-related changes of gut microbiota composition and functional profiles after 4 months of weight loss intervention. Eur J Nutr. 2021 Sep;60(6):3279-3301. doi: 10.1007/s00394-021-02508-0. Epub 2021 Feb 16. PMID 33591390
- [Derived] Ramos-Lopez O, Cuervo M, Goni L, Milagro FI, Riezu-Boj JI, Martinez JA. Modeling of an integrative prototype based on genetic, phenotypic, and environmental information for personalized prescription of energy-restricted diets in overweight/obese subjects. Am J Clin Nutr. 2020 Feb 1;111(2):459-470. doi: 10.1093/ajcn/nqz286. PMID 31751449
- [Derived] Ramos-Lopez O, Riezu-Boj JI, Milagro FI, Goni L, Cuervo M, Martinez JA. Differential lipid metabolism outcomes associated with ADRB2 gene polymorphisms in response to two dietary interventions in overweight/obese subjects. Nutr Metab Cardiovasc Dis. 2018 Feb;28(2):165-172. doi: 10.1016/j.numecd.2017.11.006. Epub 2017 Dec 5. PMID 29331538